CLINICAL TRIAL: NCT02990130
Title: Biochemical and Physiologic Factors That Affect Patient Fitness and Body Composition During Hematopoietic Stem Cell Transplantation for Hematologic Malignancies
Brief Title: Patient Fitness and Body Composition During Hematopoietic Stem Cell Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Garcia, Jose M., MD, PhD (Individual)
Responsible Party: Sponsor
Other Study IDs: 00935
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: This is a pilot observational study involving patients enrolled in the Seattle VA Bone Marrow Transplant Unit (BMTU) for treatment of their hematologic malignancy. Measurements of patient fitness, body composition, and inflammatory milieu will be performed at visits before HCT, and 30 days (+/- 10 days) after HCT. For patients that continue to receive care at the Seattle VA, additional visits (not exceeding 6 total) may be requested periodically for up to 2 years after HCT.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
This proposal aims to characterize biochemical and physiologic factors that contribute to changes in patient fitness and body composition during hematopoietic stem cell transplantation (HCT) for hematologic malignancies. The study group will consist of 60 patients with hematologic malignancies treated with HCT. Measurements of patient fitness, body composition, and inflammatory milieu will be performed at visits before HCT, and 30 days (+/- 10 days) after HCT. For patients that continue to receive care at the Seattle VA, additional visits (not exceeding 6 total) may be requested periodically for up to 2 years after HCT.

DETAILED DESCRIPTION:
This proposal aims to characterize biochemical and physiologic factors that contribute to changes in patient fitness and body composition during hematopoietic stem cell transplantation (HCT) for hematologic malignancies. The investigators hypothesize that: 1) HCT for hematologic malignancies is associated with a change in biochemical and physiologic factors that reflect patient fitness and 2) Baseline (pre-HCT) and post-HCT changes of biochemical and physiologic factors that reflect patient fitness are associated with HCT-related clinical outcomes.This is a pilot study involving patients enrolled in the Seattle VA Bone Marrow Transplant Unit (BMTU) for treatment of their hematologic malignancy. No vulnerable population will be included. The study group will consist of 60 patients with hematologic malignancies treated with HCT.

Measurements of patient fitness, body composition, and inflammatory milieu will be performed at visits before HCT, and 30 days (+/- 10 days) after HCT. For patients that continue to receive care at the Seattle VA, additional visits (not exceeding 6 total) may be requested periodically for up to 2 years after HCT. Data collection may include:

1. Blood tests other than those performed as clinical standard of care may include: anabolic and catabolic factors such as IGF-1, GH, IGFBP-3, free and weakly bound testosterone, IL-6, CRP, TNF-alpha, and pre-albumin.
2. Measurements of fitness other than those obtained as clinical standard of care may include: resting energy expenditure (REE) assessed by indirect calorimetry; body composition measured by bio-impedance (BIA) and dual-energy x-ray absorptiometry (DEXA) scan; handgrip strength; stair climbing power; 6-minute walk test; muscle strength; maximal oxygen consumption (VO2 max); and previously validated questionnaires to assess patient quality of life (QOL) and functional status.
3. Additional data that may be collected for this protocol will include clinical and laboratory data acquired per standard of clinical care as pertains to subjects' co-morbidities, hematologic disease and treatment history, and clinical course including nutritional status, use of nutrition support, and estimated nutritional requirements per routine dietitian assessments. A Food Frequency Questionnaire will be administered by a dietitian in addition to the routine clinical assessments.

The primary endpoint of this study is the change over time of patient fitness as assessed by the 6 minute walk test through HCT. Secondary endpoints will include other markers of anabolism and catabolism, and data collected as mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hematologic malignancy.
* Undergoing evaluation at the BMTU at the Puget Sound VA.
* Planning or receiving an autologous or allogeneic HCT

Exclusion Criteria:

• Patients who for any reason elect not to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will consist of 60 patients with hematologic malignancies treated with HCT
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-12 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test change | from baseline to 30 days (+/- 10 days) after HCT
  maximum distance walked in 6 minutes

SECONDARY OUTCOMES:
Anabolic marker changes | from baseline to 30 days (+/- 10 days) after HCT
  IGF-1, GH, IGFBP-3, free and weakly bound testosterone
Inflammatory marker changes | from baseline to 30 days (+/- 10 days) after HCT
  IL-6, CRP, TNF-alpha, and pre-albumin
Muscle strength | from baseline to 30 days (+/- 10 days) after HCT
  handgrip strength; 1-RM
resting energy expenditure changes | from baseline to 30 days (+/- 10 days) after HCT
  indirect calorimetry
body composition changes | from baseline to 30 days (+/- 10 days) after HCT
  bio-impedance and dual-energy x-ray absorptiometry (all in kg)
physical function changes | from baseline to 30 days (+/- 10 days) after HCT
  stair climbing power
maximal oxygen consumption changes | from baseline to 30 days (+/- 10 days) after HCT
  VO2 max
Quality of Life change score | from baseline to 30 days (+/- 10 days) after HCT
  ASAS
Quality of Life change score | from baseline to 30 days (+/- 10 days) after HCT
  FACIT
Quality of Life change score | from baseline to 30 days (+/- 10 days) after HCT
  Karnofsky
Quality of Life change score | from baseline to 30 days (+/- 10 days) after HCT
  ECOG
Food Frequency Questionnaire | from baseline to 30 days (+/- 10 days) after HCT
nutritional status | from baseline to 30 days (+/- 10 days) after HCT
use of nutrition support | from baseline to 30 days (+/- 10 days) after HCT
estimated nutritional requirements | from baseline to 30 days (+/- 10 days) after HCT

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No